CLINICAL TRIAL: NCT07056309
Title: A Study on Pharmacokinetics of Remternetug Administered Subcutaneously Through an Autoinjector Versus Prefilled Syringe in Healthy Participants
Brief Title: A Study of Remternetug (LY3372993) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18471; J1G-MC-LAKG (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-06-24; First posted 2025-07-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remternetug (Test) (Experimental): Remternetug administered subcutaneously (SC) via autoinjector (AI)
  Interventions: Drug: Remternetug (Test)
- Remternetug (Reference) (Experimental): Remternetug administered SC via prefilled syringe.
  Interventions: Drug: Remternetug (Reference)

INTERVENTIONS:
Drug: Remternetug (Test) — Administered SC
  Other Names: LY3372993
  Arms: Remternetug (Test)
Drug: Remternetug (Reference) — Administered SC
  Other Names: LY3372993
  Arms: Remternetug (Reference)

SUMMARY:
The main purpose of this study is to evaluate to different formulations of remternetug after single subcutaneous (SC) administration with either an autoinjector (AI) or a prefilled syringe (PFS). The study will look at the amount of remternetug that gets into the bloodstream and how long it takes the body to get rid of the remternetug when given as two different formulations.

Participation in the study will last approximately 155 days.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Have a body mass index within the range of 18.0 to 34.0 kilograms per meter squared (kg/m2) (inclusive).

Exclusion Criteria:

* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs or of constituting a risk when taking the study drug or of interfering with the interpretation of data.
* Have evidence of significant active neuropsychiatric disease, as determined by the investigator.
* Have a personal or family history of early onset AD (AD diagnosed prior to 65 years of age).
* Contraindication to MRI, including claustrophobia that cannot be managed with low-dose sedatives or the presence of contraindicated metal (ferromagnetic) implants/cardiac pacemakers.
* Intend to use over-the-counter or prescription medication, including herbal medications and traditional medications, with the exception of vitamin/mineral supplements, any hormone replacement therapy, and/or thyroid replacement therapy, within 7 days prior to dosing and for the duration of the study.
* Have a brain MRI that demonstrates any clinically significant findings that, in the opinion of the investigator, may impact the participant's ability to safely participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK): Maximum Concentration (Cmax) of Remternetug | Predose up to Day 85
Pharmacokinetic (PK): Area Under the Concentration Versus Time Curve from Zero to time t [AUC(0-t)] of Remternetug | Predose up to Day 85
Pharmacokinetic (PK): Area Under the Concentration Versus Time Curve from Zero to Infinity [AUC(0-inf)] of Remternetug | Predose up to Day 85

SECONDARY OUTCOMES:
Pharmacokinetic (PK): Time of Maximum Concentration (tmax) of Remternetug | Predose up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - QPS Missouri, Springfield, Missouri
  - Fortrea Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No